CLINICAL TRIAL: NCT05395208
Title: The Effect Of Whıte Noıse Therapeutıc Touch On Paın Level And Physıologıcal Parameters In Perıpheral Iv Catheter Interactıon In Premature Infants
Brief Title: The Effect Of White Noise And Therapeutic Touch On Pain And Physiological Parameters In Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Zeynep Uysal, NURSE, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/99
Record Dates: First submitted 2022-05-12; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled two groups (control groups and intervention group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic touch group accompanied by white noise (Experimental): * Camera recording was started 5 minutes before intravenous catheter intervention, vital signs and pain were evaluated.
  * Therapeutic touch application with white noise was started.
  * Vital signs and pain were evaluated during intravenous catheterization.
  * Vital signs and pain were evaluated when the intravenous catheter intervention was terminated and 5 minutes later, and the camera recording was stopped.
  Interventions: Behavioral: Therapeutic touch group accompanied by white noise
- Control group (No Intervention): * Camera recording was started 5 minutes before the intravenous catheter intervention, vital signs and pain were evaluated.
  * No application was made other than intravascular catheter intervention.
  * Vital signs and pain were evaluated during intravenous catheterization.
  * Vital signs and pain were evaluated when the intravenous catheter intervention was terminated and 5 minutes later, and the camera recording was stopped.

INTERVENTIONS:
Behavioral: Therapeutic touch group accompanied by white noise — During the intravenous catheter intervention, approximately 15-20 minutes of white noise was applied with therapeutic touch.
  Arms: Therapeutic touch group accompanied by white noise

SUMMARY:
Newborns hospitalized with some respiratory problems in the clinic are taken to noninvasive mechanical ventilation support and vascular access is required for some treatments to be applied to these newborns. The presence of nasal cannulas used for noninvasive mechanical ventilation support in newborns causes restlessness, agitation and stress in infants. The uneasiness and stress experienced by babies during vascular access also affects effective vascular access, causing other doses to be delayed or skipped due to treatment doses that are not completed on time. In addition, the pain experienced by babies indirectly affects nurses. It has been reported in many studies that it is effective in reducing the pain experienced by newborns with non-pharmacological methods. Simultaneous white noise will be played and therapeutic touch applied to help touch methods and white noise listening help reduce or control newborns' pain. Many studies have shown that touching to and listening white noise is effective in reducing pain. This study was planned as a randomized controlled experimental study to determine the effect of white noise-accompanied therapeutic touch application on pain level and physiological parameters and noninvasive mechanical ventilation support during peripheral intravenous catheterization in premature infants hospitalized for treatment.

Hypothesis 0: The application of therapeutic touch with white noise during peripheral intravenous catheter intervention in premature infants has no effect on the level of pain.

Hypothesis 1: White noise-accompanied therapeutic touch application reduces pain level during peripheral intravenous catheter intervention in premature infants.

Hypothesis 2: The therapeutic touch application accompanied by white noise during peripheral intravenous catheter intervention in premature infants positively affects physiological parameters.

DETAILED DESCRIPTION:
Purpose of the research The study was planned as a randomized controlled experimental study to determine the effect of white noise and therapeutic touch on pain level and physiological parameters and noninvasive mechanical ventilation support during peripheral intravenous catheter intervention in hospitalized premature infants.

As a data collection tool; "Baby Follow-up Form" was used in which some descriptive features of the baby and NIPS and physiological parameter measurements were evaluated.

Application:

The data of the study were collected using simple random sampling method. The newborns to be included in the study were divided into two groups as the intervention group and the control group. The data were determined according to the odd and even numbered days of the calendar between the research dates, and the babies born on the odd numbered days of the calendar were included in the white noise therapeutic touch group (intervention group), and the babies born on the even numbered days of the calendar were included in the control group. The environmental conditions in the two groups were regulated in the same way. The application was carried out with a research nurse performing therapeutic touch, an observer nurse and a practitioner nurse.

Intervention Group (n=40) :

* Camera recording was started 5 minutes before intravenous catheter intervention, vital signs and pain were evaluated.
* Therapeutic touch application with white noise was started.
* Vital signs and pain were evaluated during intravenous catheterization.
* Vital signs and pain were evaluated when the intravenous catheter intervention was terminated and 5 minutes later, and the camera recording was stopped.

Control Group (n=41):

* Camera recording was started 5 minutes before the intravenous catheter intervention, vital signs and pain were evaluated.
* No application was made other than intravascular catheter intervention.
* Vital signs and pain were evaluated during intravenous catheterization.
* Vital signs and pain were evaluated when the intravenous catheter intervention was terminated and 5 minutes later, and the camera recording was stopped.

Universe and Research Example Newborns treated at Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital Neonatal Intensive Care Service between June 2021 and January 2022 constitute the population of the research. The sample of the study consisted of 85 newborns meeting the sampling criteria of the study in the Neonatal Intensive Care Service of Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital.

Sampling selection criteria of the infant;

* 32-36. to be born in gestational weeks,
* The need for noninvasive mechanical ventilation,
* Absence of congenital anomalies,
* Appropriate cognitive level and motor development of the newborn,
* Does not prevent the opening of the vascular access,
* Not using narcotic, sedative opioid and anticonvulsant drugs,
* No pharmacological intervention for the baby's pain during the procedure,
* Parents sign the informed consent form. Dependent Variables: The newborn's heart rate, respiratory rate, oxygen saturation, body temperature, blood pressure, pain score are the dependent variables.

Independent Variables: The sex of the newborn, gestational age, mode of delivery, weight, height, head circumference, type of feeding, type of noninvasive mechanical ventilation support constitute the independent variables.

Sample size was determined by power analysis. In the study, the power of the sample was calculated with the G*Power 3.1 program. The amount of type I error was 0.05 and the power of the test =0.80 (α=0.05, 1-β=0.80, effect size:0.6), while the minimum sample size (36 newborns in each group) was 72. newborns Considering the losses that may arise from the sample for any reason during the study period, it is planned to take 10% more of the power analysis result. In the study, 40 newborns were included in the intervention group (therapeutic touch with white noise) and 41 newborns in the control group.

Data Collection Written permission from the ethics committee of Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital (Annex-3) and research permission from the Istanbul Governorship Provincial Health Directorate (Annex-4) for the collection of pre-research data. After explanations were given to the families of the newborns who agreed to participate in the study, and to the families of the newborns who met the sample selection criteria for the purpose of the study, verbal and written informed consent was obtained from the families of the newborns who agreed to participate in the study (Annex-1). During the research, personal information will be kept confidential and care will be taken for their privacy. The data of the study were collected between June 2020 and January 2021. The application time of each data and filling the data collection forms took an average of 20-25 minutes.

Evaluation of Data The data of the study were analyzed with appropriate statistical methods using the SPSS (Statistical Package for the Social Science) 22.0 package program. In the evaluation of the data, percentage, number, mean and standard deviation were used as descriptive statistical methods, and frequency and percentage distributions of the data were given. The relationship between the variables measured at the categorical level was evaluated with the Pearson chi-square test. Whether the research variables showed normal distribution or not was examined by paired test and independent group t test. The significance level was 0.05; It was stated that there was a significant difference in cases with p<0.05, and there was no significant difference in cases with p>0.05.

ELIGIBILITY:
Inclusion Criteria:

* To be in noninvasive mechanical ventilation support,
* Newborns between 32-36 weeks,
* Not having a life-threatening disease,
* No congenital anomalies,
* Appropriate cognitive level and motor development of the newborn,
* The newborn does not have a physical problem,
* Parents' willingness to participate in the research,

Exclusion Criteria:

* Presence of IV catheter,
* Having a condition that prevents vascular access,
* Those who have circulation problems in the body,
* Using narcotic, sedative opioid and anticonvulsant drugs
* Pharmacological intervention application for the baby's pain during the procedure

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Pain Score | Before intravenous catheter intervention (5 minutes ago)
  NIPS: Newborn Infant Pain Scale was evaluated. The Newborn Infant Pain Scale consists of 6 behavioral parts: facial expression, crying, breathing pattern, arm and leg movements, and alertness. Apart from crying, 2 separate points (0-1 points) are given for other behaviors, and 3 separate points (0-1-2) are given for crying. The total score varies between 0-7. A high score indicates increased pain intensity. According to the scale scoring: 0 Points: No pain, 1-2 Points: Mild pain, 3-4 Points: Moderate pain, 5-7 Points: Severe pain.
Pain Score | Intravenous catheter attempt sequence (0th. minute)
  NIPS: Newborn Infant Pain Scale was evaluated. The Newborn Infant Pain Scale consists of 6 behavioral parts: facial expression, crying, breathing pattern, arm and leg movements, and alertness. Apart from crying, 2 separate points (0-1 points) are given for other behaviors, and 3 separate points (0-1-2) are given for crying. The total score varies between 0-7. A high score indicates increased pain intensity. According to the scale scoring: 0 Points: No pain, 1-2 Points: Mild pain, 3-4 Points: Moderate pain, 5-7 Points: Severe pain.
Pain Score | Immediately after intravenous catheter intervention (0th minute)
  NIPS: Newborn Infant Pain Scale was evaluated. The Newborn Infant Pain Scale consists of 6 behavioral parts: facial expression, crying, breathing pattern, arm and leg movements, and alertness. Apart from crying, 2 separate points (0-1 points) are given for other behaviors, and 3 separate points (0-1-2) are given for crying. The total score varies between 0-7. A high score indicates increased pain intensity. According to the scale scoring: 0 Points: No pain, 1-2 Points: Mild pain, 3-4 Points: Moderate pain, 5-7 Points: Severe pain.
Pain Score | 5 minutes after intravenous catheterization
  NIPS: Newborn Infant Pain Scale was evaluated. The Newborn Infant Pain Scale consists of 6 behavioral parts: facial expression, crying, breathing pattern, arm and leg movements, and alertness. Apart from crying, 2 separate points (0-1 points) are given for other behaviors, and 3 separate points (0-1-2) are given for crying. The total score varies between 0-7. A high score indicates increased pain intensity. According to the scale scoring: 0 Points: No pain, 1-2 Points: Mild pain, 3-4 Points: Moderate pain, 5-7 Points: Severe pain.

SECONDARY OUTCOMES:
Blood pressure Vital Signs | Before intravenous catheter intervention (5 minutes ago)
  Blood pressure (mmHg) were evaluated
Blood pressure Vital Signs | Immediately after intravenous catheter intervention (0th minute)
  Blood pressure (mmHg) were evaluated
Blood pressure Vital Signs | 5 minutes after intravenous catheterization
  Blood pressure (mmHg) were evaluated
Oxygen saturation Vital Signs | Before intravenous catheter intervention (5 minutes ago)
  Oxygen saturation (%) were evaluated
Oxygen saturation Vital Signs | Intravenous catheter attempt sequence (0th. minute)
  Oxygen saturation (%) were evaluated
Oxygen saturation Vital Signs | Immediately after intravenous catheter intervention (0th minute)
  Oxygen saturation (%) were evaluated
Oxygen saturation Vital Signs | 5 minutes after intravenous catheterization
  Oxygen saturation (%) were evaluated
Heart rate Vital Signs | Before intravenous catheter intervention (5 minutes ago)
  Heart rate (beats/minute) were evaluated
Heart rate Vital Signs | Intravenous catheter attempt sequence (0th. minute)
  Heart rate (beats/minute) were evaluated
Heart rate Vital Signs | Immediately after intravenous catheter intervention (0th minute)
  Heart rate (beats/minute) were evaluated
Heart rate Vital Signs | 5 minutes after intravenous catheterization
  Heart rate (beats/minute) were evaluated
Respiratory Rate Vital Signs | Before intravenous catheter intervention (5 minutes ago)
  Respiratory Rate (breaths/minute) were evaluated
Respiratory Rate Vital Signs | Intravenous catheter attempt sequence (0th. minute)
  Respiratory Rate (breaths/minute) were evaluated
Respiratory Rate Vital Signs | Immediately after intravenous catheter intervention (0th minute)
  Respiratory Rate (breaths/minute) were evaluated
Respiratory Rate Vital Signs | 5 minutes after intravenous catheterization
  Respiratory Rate (breaths/minute) were evaluated
Body temperature Vital Signs | Before intravenous catheter intervention (5 minutes ago)
  Body temperature (°C) were evaluated
Body temperature Vital Signs | Intravenous catheter attempt sequence (0th. minute)
  Body temperature (°C) were evaluated
Body temperature Vital Signs | Immediately after intravenous catheter intervention (0th minute)
  Body temperature (°C) were evaluated
Body temperature Vital Signs | 5 minutes after intravenous catheterization
  Body temperature (°C) were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Gülzade Uysal, Assoc. Dr., Study Director — Okan Üniversitesi
Locations (1):
- Home/Work, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No